CLINICAL TRIAL: NCT00213941
Title: Study Protocol Evaluating Transient Tachypnoea of the Newborn in Term and Near Term Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3214
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-10

CONDITIONS: Transient Tachypnoea of the Newborn
Keywords: transient tachypnoea of the newborn; surfactant deficiency; persistant pulmonary hypertension of the neonate; lung maturity tests
MeSH Terms: conditions — Transient Tachypnea of the Newborn | interventions — Echocardiography

INTERVENTIONS:
Device: Echocardiography

SUMMARY:
Transient tachypnoea of the newborn (TTN) is a common cause of hospitalisation in the neonatal period, complicating 1 to 1,5 per cent life birth. Predisposing factors are prematurity, birth after C section, especially before the onset of labor. The main factor leading to this condition is a lack of absorption of the fluid contained in the alveolar space resulting in an early respiratory distress which normally resolves in two to five days with oxygen supplementation.

Meanwhile, some neonates will experience a complicated evolution requiring ventilatory support and hospitalisatioon in neonatal intensive care unit. This complication is not preventable and could result either of a surfactant deficiency (primary or secondary) or a persistent pulmonary hypertension of the neonate (PPHN).

In this study, a cohort of newborn presenting TTN will be followed, in order to evaluate, at initial admission, pulmonary maturation (with fetal lung maturity test and the stable microbubble test) and to seek for PPHN (echochardiography). Therapeutic management will be done according to standard care and classification of the neonate will be performed according to their clinical evolution: group 1 (uncomplicated TTN) and group 2 (complicated TTN).

Statistical analysis will compare results of the tests at initial evaluation in the two groups, and accuracy of the tests to predict a complicated evolution will be established.

ELIGIBILITY:
Inclusion Criteria:

* Neonate > or = 34 weeks GA admitted in the first 6 hours of life with the suspected diagnosis of TTN (respiratory rate > 60/mn, SpO2 < 90% in room air, ilvermann score > 0
* Parental consent obtained

Exclusion Criteria:

* GA> 42 weeks
* meconial amniotic fluid
* early onset neonatal sepsis (septic shock)
* congenital malformations
* enteral feeding started before admission
* no parental consent

Ages: 0 Years to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2004-11

PRIMARY OUTCOMES:
Evaluate and compare the accuracy of different tests at initial evaluation in predicting a complicated course in neonae with TTN

SECONDARY OUTCOMES:
Increase the knowledge in the physiopathology of TTN

CONTACTS AND LOCATIONS:
Overall Officials: Pierre KUHN, MD, Principal Investigator — Service de Pédiatrie, Hôpital de Hautepierre
Locations (1):
- Service de Pédiatrie 2, Hôpital de Hautepierre, Strasbourg, France